CLINICAL TRIAL: NCT06365541
Title: Exploring the Efficacy and Safety of Dapagliflozin in Improving Heart Failure in Dialysis Patients: an Open, Prospective, and Self-controlled Study
Brief Title: The Efficacy and Safety of Dapagliflozin in Improving Heart Failure in Dialysis Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The People's Hospital of Gaozhou (Other)
Responsible Party: Principal Investigator, deng shanshan, Researcher, The People's Hospital of Gaozhou
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GYLLPJ-2024006
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: The Efficacy and Safety of Dapagliflozin in Improving Heart Failure in Dialysis Patients
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Exploring the efficacy and safety of dapagliflozin in improving heart failure in dialysis patients by the analysis and comparison of patients' own data before and after dapagliflozin treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self Control (Experimental): Compare the heart function of dialysis patients before treatment and during the third and sixth months of treatment.
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — oral Dapagliflozin tablets 10mg/day for 6 months

SUMMARY:
Dialysis patients have a higher incidence of cardiovascular events and require more effective measures to delay the progression of heart failure. Many studies have shown that dapagliflozin has cardioprotective effect, but most studies focus on non-dialysis patients with eGFR more than 20ml/min/1.73m2. However, the data on patients with eGFR less than 20ml/min/1.73m2 or dialysis patients, especially peritoneal dialysis patients, is less. Exploring the efficacy and safety of Dapagliflozin in improving heart failure in dialysis patients is of great clinical significance.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age between 20 and 70 years old; 2.Maintenance dialysis for longer than 3 months; 3.Diagnosis with chronic heart failure, Left ventricular ejection fraction (LVEF)≤40% or NT-proBNP>12000pg/ml; 4.The patient signs an informed consent form.

Exclusion Criteria:

* 1.Patients with liver function impairment; 2.Patients with severe hypoglycemia/hypotension/ketoacidosis; 3.Patients with active pyelonephritis or symptomatic urinary tract infection; 4.Dapagliflozin allergies or severe adverse reactions; 5.Patients suffering from other severe diseases; 6.Patients participating in other clinical trials; 7.Pregnant or lactating women; 8.Failure to sign a written informed consent form; 9.Unable or unwilling to comply with the experimental protocol approved by the researcher

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
N-terminal B-type natriuretic peptide precursor (NT-proBNP) | Baseline, 3 months, 6 months
  Changes in NT-proBNP levels before and after treatment
Left ventricular ejection fraction (LVEF) | Baseline, 3 months, 6 months
  Changes in LVEF levels before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The People's Hospital of Gaozhou, Maoming, Guangdong, China

IPD SHARING:
Plan to Share IPD: No